CLINICAL TRIAL: NCT03131037
Title: Intratumoral Gene Mediated Cytotoxic Immunotherapy (GMCI) For Resectable Non-Small Cell Lung Cancer
Brief Title: Intratumoral Gene Mediated Cytotoxic Immunotherapy in Patients With Resectable Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuTK01
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
Keywords: aglatimagene besadenovec; CAN-2409; immunotherapy; GMCI; AdV-tk
MeSH Terms: conditions — Lung Neoplasms | interventions — Valacyclovir

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): CAN-2409 + valacyclovir
  Interventions: Biological: CAN-2409 + valacyclovir

INTERVENTIONS:
Biological: CAN-2409 + valacyclovir — CAN-2409 will be administered intratumorally followed by oral valacyclovir. Valacyclovir will be administered orally at a fixed dose for 14 days after each injection.

SUMMARY:
This is a phase I dose escalation study of CAN-2409 plus prodrug in patients with non-small cell lung cancer (NSCLC). The primary clinical objective of the study is to evaluate the safety of CAN-2409 plus prodrug when combined with standard surgery for NSCLC. The primary scientific objective is to determine the immunologic changes induced by CAN-2409 plus prodrug.

DETAILED DESCRIPTION:
The purpose of this open-label, dose escalation clinical trial is to investigate the safety of CAN-2409 (aglatimagene besadenovec) plus prodrug prior to surgery in patients with NSCLC. CAN-2409 is a viral immunotherapy approach which utilizes intratumoral administration to selectively induce tumor cell death and elicit both an innate and an adaptive systemic anti-tumor immune response against the injected tumor and uninjected metastases. Local delivery enables these effects while aiming to minimize systemic toxicity. Standard of care surgical resection will be performed about 3 weeks after the CAN-2409 injection. Chemotherapy and/or radiation may begin 6-8 weeks after resection surgery. Choice of chemotherapy depends on the treating oncologist. CAN-2409 (aglatimagene besadenovec) was previously known as AdV-tk, and the combination of CAN-2409 plus prodrug was previously known as GMCI.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented non-small cell carcinoma (cytology or histology) that is accessible via standard-of-care staging procedures: (1) EBUS or (2) surgical approaches (eg mediastinoscopy, mediastinotomy or VATS).
* Resectable with negative lymph nodes based on imaging with histologic confirmation at time of the staging procedure prior to AdV-tk injection
* The tumor must be 4cm or greater in diameter based on imaging
* ECOG Performance status of 0 or 1.
* Granulocyte count (ANC) ≥ 1,000/mm3
* Peripheral lymphocyte count ≥ 500/mm3
* Hemoglobin ≥ 9 g/dl
* Platelets ≥ 100,000/mm3
* Total bilirubin ≤ 1.5 x upper limit of normal
* SGOT (AST) ≤ 3x upper limit of normal
* Serum creatinine < 2mg/dl
* Calculated creatinine clearance > 30ml/min
* Patients must give study specific informed consent prior to enrollment

Exclusion Criteria:

* Radiotherapy and/or treatment with chemotherapeutic, cytotoxic, or immunologic agents within 4 weeks prior to infusion of the vector.
* Known immunodeficiency such as HIV infection
* Active liver disease, including known cirrhosis or active hepatitis
* Use of systemic corticosteroids (>10 mg prednisone per day or equivalent) or other systemic immunosuppressive drugs
* Patient is pregnant or breast-feeding. Female patients of childbearing age must have negative serum or urine pregnancy test within 1 week of beginning therapy. Subjects must use acceptable means of birth control until 30 days after the vector injection.
* Presence of any other life-threatening illness, such as unstable angina, severe oxygen dependence, significant chronic obstructive pulmonary disease (COPD), end-stage liver or renal disease. COPD will be considered significant if disease limits activities of daily living, results in the inability to walk up 1 flight of stair, or requires home oxygen.
* Presence of known untreated brain metastases.
* Prior bone marrow transplants (including stem cells) except autologous stem cell transplant without immunosuppression is NOT considered an exclusion.
* Known sensitivity or allergic reactions to valacyclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 6 weeks

SECONDARY OUTCOMES:
Progression free survival (PFS) | 5 years
Overall survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Predina JD, Haas AR, Martinez M, O'Brien S, Moon EK, Woodruff P, Stadanlick J, Corbett C, Frenzel-Sulyok L, Bryski MG, Eruslanov E, Deshpande C, Langer C, Aguilar LK, Guzik BW, Manzanera AG, Aguilar-Cordova E, Singhal S, Albelda SM. Neoadjuvant Gene-Mediated Cytotoxic Immunotherapy for Non-Small-Cell Lung Cancer: Safety and Immunologic Activity. Mol Ther. 2021 Feb 3;29(2):658-670. doi: 10.1016/j.ymthe.2020.11.001. Epub 2020 Nov 5. PMID 33160076
- See also: Neoadjuvant Gene-Mediated Cytotoxic Immunotherapy for Non-Small-Cell Lung Cancer: Safety and Immunologic Activity — https://pubmed.ncbi.nlm.nih.gov/33160076/